CLINICAL TRIAL: NCT04960514
Title: A Prospective Decision Impact Trial of KidneyIntelX in Patients With Type 2 Diabetes and Existing Chronic Kidney Disease
Brief Title: Prospective Decision Impact Trial of KidneyIntelX
Status: Active, not recruiting | Type: Observational
Sponsor: Renalytix AI, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RAI 19-1003
Record Dates: First submitted 2021-07-02; First posted 2021-07-14 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Kidney Disease; Chronic Kidney Disease Stage 1; Chronic Kidney Disease Stage 2; Chronic Kidney Disease, Stage 3 (Moderate)
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: KidneyIntelX — KidneyIntelX is a blood-based clinical diagnostic tool that assesses the risk of progressive kidney function decline in chronic kidney disease patients with type 2 diabetes.

SUMMARY:
The current trial is designed to evaluate how the results of KidneyIntelX test / platform impacts on the clinical management of type 2 diabetes patients identified as increased risk for rapid kidney function decline within 5-years.

ELIGIBILITY:
Inclusion Criteria:

* 23 years of age or older.
* Clinical history of confirmed type 2 diabetes.
* Evidence of DKD Stages 1-3:
* Baseline eGFR of 30-59 ml/min/1.73m2 (confirmed 3 months apart with at least one value within 1 year prior to enrollment)
* Individuals with eGFR ≥60 ml/min/1.73m2 and albuminuria (UACR ≥30mg/g)
* All patients will have a HbA1c, eGFR, urine albumin and urine creatinine, eGFR, available from within 12 months of enrollment (to be obtained if not clinically available prior).
* The subject must be able to comprehend and sign an approved informed consent form and other applicable study documents.

Exclusion Criteria:

* Patients with eGFR <30 or ≥ 60 ml/min/1.73m2 without albuminuria.
* Patients with ESRD or on renal recovery treatments at time of enrollment.
* Patients who are pregnant at the time of enrollment.
* Patients who are currently hospitalized.
* Patients who are currently on Enbrel.

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 diabetes and existing chronic kidney disease stages 1-3.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 12 Months
  Proportion (target: 20% increase from prior measurements) of visits in which each participant achieves target blood pressure of <140/90 mmHg (as per the NKF CKD management guidelines).
HbA1c | 12 Months
  Proportion (target: 20% increase) of patients that achieve individualized target of HbA1c.
ACEi/ARB | 12 Months
  Proportion (target: 20% increase) of patients recently treated with statins and or angiotensin-converting-enzyme inhibitors and angiotensin II receptor blockers.
SGLT2/ GLP1 | 12 Months
  Proportion (target: 20% increase) of patients recently treated with SGLT2 inhibitors or GLP1 agonists.
Urine albumin to creatinine ratio | 12 Months
  In those with baseline albuminuria, proportion (target: 20%) of patients achieving a 30% decrease in their urine albumin to creatinine ratio from averaged pre-enrollment values to average post-enrollment values through 1 year.
Referrals | 12 Months
  Proportion (target: 20% increase) of patients referred/managed by a dietician, diabetologist, or nephrologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Atrium Health Wake Forest Baptist - Family Medicine - Piedmont Plaza, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided